CLINICAL TRIAL: NCT06538818
Title: Ultra Phonophoresis With a Hyaluronic Acid-Containing Gel on Carpal Tunnel Syndrome Related Hormonal Therapy Post Mastectomy.
Brief Title: Ultra Phonophoresis With a Hyaluronic Acid-Containing Gel on Carpal Tunnel Syndrome Post Mastectomy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Gamal Fawzy El-Sayed, Lecturer of physical therapy of surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005219
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Mastectomy; Carpal Tunnel Syndrome (CTS)
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Experimental): This group will include 30 patients who will receive Ultra Phonophoresis with a hyaluronic acid-containing gel 5 sessions per week for 3 weeks in addition to their physical therapy program and medical treatment.
  Interventions: Device: Ultra Phonophoresis
- Control group: (No Intervention): This group will include 30 patients who will receive only their traditional physical therapy program and medical treatment.

INTERVENTIONS:
Device: Ultra Phonophoresis — Therapeutic pulsed ultrasound using Phyaction UbMF ultrasound device in presence of a hyaluronic acid-containing gel will be applied gel pad over the wrist and along the course of median nerve at the carpal tunnel.
  The following parameters will be used: intensity of 1.0 W/em2 at a 1MHz frequency for 5 minutes and pulsed (25%) ultrasound waves to transfer the hyaluronic acid-containing gel. This therapy will be applied for 5 min/session, 5 d/wk, for 3 weeks.
  The following parameters will be used:
  * intensity of 1.0 W/cm2
  * 1MHz frequency
  * pulsed (25%)
  * 5 min/session, 5 d/wk, for 3 weeks.
  Arms: Study group

SUMMARY:
In this study, 60 patients will be randomly assigned into two equal groups (30 patients for each group):

1. Group A: This group will include 30 patients who will receive Ultra Phonophoresis with a hyaluronic acid-containing gel 5 sessions per week for 3 weeks in addition to their physical therapy program and medical treatment.
2. Group B: This group will include 30 patients who will receive only their traditional physical therapy program and medical treatment.

Criteria for the patient selection:

(A) Inclusion Criteria:

The subject selection will be according to the following criteria:

* Age range between 40-55 years.
* Female patients will participate in the study.
* All patients will have hormonal therapy at least for 6 weeks.
* All patients enrolled to the study will have their informed consent.
* Patient referred from physician by carpal tunnel syndrome. (B) Exclusion Criteria:

The potential participants will be excluded if they meet one of the following criteria:

* Marked lymphedema.
* Steroid injection for CTS.
* Thrombosis propensity.
* Cervical radiculopathy.
* Brachial plexopathy

DETAILED DESCRIPTION:
1. Assessment measures and procedures:

   The outcome measures will include Median nerve sensory and motor distal latency, arm volume calculated by circumference measurement, pain using a visual analogue scale (VAS) and Boston Carpal Tunnel Questionnaire (BCTQ). Assessment will conducted by a physiotherapist pre-and post-treatment.
   1. Nerve conduction studies:

      Electro diagnostic assessment will conducted by a physical medicine specialist. During the study, the temperature of patients' hands will be kept >32. For assessing the Motor distal latency, the active recording electrode will be fastened on abductor pollicis brevis (APB) muscle and median nerve will be stimulated at wrist region with stimulator electrode, 8 cm proximal to the active electrode and then the distal latency will be recorded. Regarding the sensory distal latency, the recorder will be fastened on the third finger, and stimulator electrode will be placed 14 cm proximal to the recorder and will stimulate median nerve once at wrist and once at palm region, then distal latency will be recorded. Normal distal sensory latency of median nerve is of less than 3.6 and distal motor latency of median nerve less than 4.2. If only the sensory distal latency will long, patient has mild CTS, but if both sensory and motor distal latency will be long and denervation will not be observed in electromyography of APB, it is moderate CTS.
   2. Visual analogue scale VAS for pain assessment:

      Intensity of pain is another outcome measure will be used to evaluate treatment. Adults use the visual analogue scale (VAS), a one-dimensional assessment tool, particularly for chronic pain. The VAS is a continuous scale that consists of a line that is either vertical (VVAS) or horizontal (HVAS), usually 10 cm long, and is supported by two verbal descriptors, one for each symptom intensity. The patients will be thoroughly briefed on the instructions, reporting timeline, and vocal description anchors prior to the measurement.
   3. Baseline hand dynamometer Baseline hydraulic hand dynamometer is used to measure hand grip strength. It is manufactured and serviced in the USA since 1978. It gives accurate grip strength readings without the subject being able to feel the handle move.

      The internationally accepted design ensures reliability, user convenience and measurement repeatability. Maximum reading remains until the unit is reset. The device comes with five position handles to improve comfort while using the dynamometer. The device Gauge is made of bourdon tube element with spring suspended movement that can viewed as pounds or kilograms.
   4. Boston Carpal Tunnel Questionnaire (BCTQ):

   Patients w Patients with CTS can assess their level of dysfunction and symptom severity using the BCTQ .It has two measurement scales: the BCTQ-F, which measures functional status, and the BCTQ-S, which measures symptom severity. The BCTQ-S employs eleven questions on a five-point rating system from 1 (no symptoms) to 5 (severe symptoms) to assess the frequency and intensity of pain, numbness, weakness, and loss of dexterity. The average scores of the 11 questions are used to analyze the results. The BCTQ-F has eight questions that are scored on a five-point scale from 1 (no trouble) to 5 (cannot do at all owing to hand or wrist symptoms) to assess the degree of difficulty in carrying out daily chores. The average scores of the eight questions are used to analyze the results.

   2-2- 50 - 100 b-Therapeutic device: a.Ultrasound device + Gel pad Phyactio n For ultrasound therapy offers a large and clear screen, with a user-friendly interface that makes it simple and easy to use. The device comes with a multi-frequency detachable head (1 / 3 MHZ and offers different pulsed and continuous modes (10 -25 - 30 - 40 - 50 - 100%).

   Device specifications:
   * -Dimensions: 265 x 275 x 122 mm
   * -Weight: 3.1 Kg
   * -Mains voltage: 100 - 240 VAC, 50/60 HZ
   * -Maximum power: 35 VA
   * -Safety class: Class I
   * -Treatment time: 0-30 minutes
2. Procedures of Ultra Phonophoresis; Therapeutic pulsed ultrasound using Phyaction UbMF ultrasound device in presence of a hyaluronic acid-containing gel will be applied gel pad over the wrist and along the course of median nerve at the carpal tunnel.

The following parameters will be used: intensity of 1.0 W/em2 at a 1MHz frequency for 5 minutes and pulsed (25%) ultrasound waves to transfer the hyaluronic acid-containing gel. This therapy will be applied for 5 min/session, 5 d/wk, for 3 weeks.

The following parameters will be used:

* intensity of 1.0 W/cm2
* 1MHz frequency
* pulsed (25%)
* 5 min/session, 5 d/wk, for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 40-55 years.
* Female patients will participate in the study.
* All patients will have hormonal therapy at least for 6 weeks.
* All patients enrolled to the study will have their informed consent.
* Patient referred from physician by carpal tunnel syndrome

Exclusion Criteria:

* -Marked lymphedema.
* Steroid injection for CTS.
* Thrombosis propensity.
* Cervical radiculopathy.
* Brachial plexopathy

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — * All patients will have hormonal therapy at least for 6 weeks.
  * Patient referred from physician by carpal tunnel syndrome post mastectomy
Enrollment: 60 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Median nerve sensory and motor distal latency | 3 weeks
  For assessing the Motor distal latency, the active recording electrode will be fastened on abductor pollicis brevis (APB) muscle and median nerve will be stimulated at wrist region with stimulator electrode, 8 cm proximal to the active electrode and then the distal latency will be recorded. Regarding the sensory distal latency, the recorder will be fastened on the third finger, and stimulator electrode will be placed 14 cm proximal to the recorder and will stimulate median nerve once at wrist and once at palm region, then distal latency will be recorded. Normal distal sensory latency of median nerve is of less than 3.6 and distal motor latency of median nerve less than 4.2. If only the sensory distal latency will long, patient has mild CTS, but if both sensory and motor distal latency will be long and denervation will not be observed in electromyography of APB, it is moderate CTS.
pain using a visual analogue scale (VAS) | 3 weeks
  Intensity of pain is another outcome measure will be used to evaluate treatment. Adults use the visual analogue scale (VAS), a one-dimensional assessment tool, particularly for chronic pain. The VAS is a continuous scale that consists of a line that is either vertical (VVAS) or horizontal (HVAS), usually 10 cm long, and is supported by two verbal descriptors, one for each symptom intensity. The patients will be thoroughly briefed on the instructions, reporting timeline, and vocal description anchors prior to the measurement.
Baseline hydraulic hand dynamometer is used to measure hand grip strength | 3 weeks
  . It is manufactured and serviced in the USA since 1978. It gives accurate grip strength readings without the subject being able to feel the handle move.
  The internationally accepted design ensures reliability, user convenience and measurement repeatability. Maximum reading remains until the unit is reset. The device comes with five position handles to improve comfort while using the dynamometer. The device Gauge is made of bourdon tube element with spring suspended movement that can viewed as pounds or kilograms.
Boston Carpal Tunnel Questionnaire (BCTQ): | 3 weeks
  Patients with CTS can assess their level of dysfunction and symptom severity using the BCTQ .It has two measurement scales: the BCTQ-F, which measures functional status, and the BCTQ-S, which measures symptom severity. The BCTQ-S employs eleven questions on a five-point rating system from 1 (no symptoms) to 5 (severe symptoms) to assess the frequency and intensity of pain, numbness, weakness, and loss of dexterity. The average scores of the 11 questions are used to analyze the results. The BCTQ-F has eight questions that are scored on a five-point scale from 1 (no trouble) to 5 (cannot do at all owing to hand or wrist symptoms) to assess the degree of difficulty in carrying out daily chores. The average scores of the eight questions are used to analyze the results.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No